CLINICAL TRIAL: NCT07390799
Title: Effect of Prophylactic Tranexamic Acid Administered After Fetal Delivery on Perioperative Blood Loss and Neonatal Outcomes in Low-Risk Repeat Cesarean Delivery: A Randomized Controlled Trial
Brief Title: Prophylactic Tranexamic Acid in Low-Risk Repeat Cesarean Delivery: A Randomized Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Sabahattin Anıl Arı, Associate Professor, Ege University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2517
Record Dates: First submitted 2026-01-29; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Cesarean Delivery
Keywords: Tranexamic Acid; Repeat Cesarean Section; Perioperative Blood Loss
MeSH Terms: interventions — Tranexamic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tranexamic Acid Group (Experimental): Participants randomized to this arm will receive a single dose of tranexamic acid (1 g) administered intravenously immediately after fetal delivery during cesarean section, in addition to standard surgical and uterotonic management.
  Interventions: Drug: Tranexamic Acid
- Control Group (No Intervention): Participants randomized to this arm will receive standard surgical and uterotonic management during cesarean section without the administration of tranexamic acid.

INTERVENTIONS:
Drug: Tranexamic Acid — Tranexamic acid 1 g will be administered intravenously as a single dose immediately after fetal delivery during cesarean section, in addition to standard surgical and uterotonic management.
  Arms: Tranexamic Acid Group

SUMMARY:
Postpartum hemorrhage remains a leading cause of maternal morbidity following cesarean delivery. Tranexamic acid (TXA) has been shown to reduce blood loss when used for the treatment of postpartum hemorrhage; however, its routine prophylactic use during cesarean delivery, particularly in low-risk women, remains controversial. Large randomized trials have demonstrated limited benefit on major maternal outcomes, and data regarding clinically meaningful blood loss reduction and neonatal safety are still inconclusive.

This randomized controlled trial aims to evaluate the effect of prophylactic tranexamic acid administered after fetal delivery on perioperative blood loss in women undergoing low-risk repeat cesarean delivery. Secondary objectives include the assessment of neonatal outcomes to further evaluate the safety of routine TXA administration in this population.

The results of this study are expected to provide evidence to inform clinical decision-making regarding the routine use of tranexamic acid in low-risk repeat cesarean deliveries, balancing potential maternal benefits against neonatal safety considerations.

DETAILED DESCRIPTION:
Postpartum hemorrhage remains one of the leading causes of maternal morbidity worldwide, and cesarean delivery is associated with a higher risk of perioperative blood loss compared with vaginal birth. Tranexamic acid (TXA), a synthetic antifibrinolytic agent, is well established for the treatment of postpartum hemorrhage. However, the role of routine prophylactic TXA administration during cesarean delivery remains controversial, particularly in women without established risk factors for excessive bleeding.

Recent large randomized trials have demonstrated that prophylactic TXA administered after fetal delivery may reduce measured blood loss but does not significantly improve major maternal outcomes such as the need for blood transfusion or maternal mortality in unselected cesarean populations. Furthermore, data regarding the clinical relevance of modest reductions in blood loss and the potential impact on neonatal outcomes remain limited.

This randomized controlled trial is designed to evaluate the effect of prophylactic tranexamic acid administered after fetal delivery on perioperative blood loss in women undergoing low-risk repeat cesarean delivery. The study focuses on women undergoing their second or third cesarean section without additional risk factors for postpartum hemorrhage, representing a clinically common yet understudied population.

Participants will be randomized in a 1:1 ratio to receive either intravenous tranexamic acid (1 g) administered immediately after fetal delivery or standard care without tranexamic acid. All participants will receive standardized surgical technique and uterotonic management according to institutional protocols. Perioperative blood loss will be measured using standardized methods. A difference of 200 mL in perioperative blood loss is considered clinically meaningful for the purposes of this study.

In addition to maternal outcomes, neonatal outcomes will be prospectively assessed to evaluate the safety of routine prophylactic TXA administration when given after fetal delivery. Neonatal assessments will include immediate postnatal adaptation, need for resuscitation, admission to the neonatal intensive care unit, and selected laboratory and clinical outcomes during the early neonatal period.

By focusing on a homogeneous low-risk repeat cesarean population and incorporating both maternal and neonatal outcomes, this study aims to clarify whether routine prophylactic tranexamic acid use provides clinically meaningful benefit without compromising neonatal safety. The findings are expected to inform evidence-based decision-making regarding the routine use of tranexamic acid in low-risk repeat cesarean delivery.

ELIGIBILITY:
Inclusion Criteria:

Women aged 18 to 45 years Singleton pregnancy Gestational age ≥37+0 weeks Scheduled second or third cesarean delivery Classified as low risk for postpartum hemorrhage Ability to provide written informed consent Planned cesarean delivery under regional or general anesthesia

Exclusion Criteria:

Primary cesarean delivery More than three previous cesarean deliveries Placenta previa, placenta accreta spectrum, or suspected abnormal placentation Multiple pregnancy Known coagulation disorders or use of anticoagulant therapy History of thromboembolic disease Severe anemia (hemoglobin <10 g/dL) Hypertensive disorders of pregnancy (including preeclampsia or eclampsia) Intrauterine fetal demise Emergency cesarean delivery Known hypersensitivity to tranexamic acid

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 204 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Perioperative blood loss (mL) | From skin incision until completion of surgery
  Perioperative blood loss will be quantified using standardized measurement methods during cesarean delivery. A difference of 200 mL in perioperative blood loss between groups is considered clinically meaningful.

CONTACTS AND LOCATIONS:
Overall Officials: Sabahattin Anıl A ARI, Associate Professor, Principal Investigator — Izmir Bakircay University
Locations (1):
- Izmir Bakircay University, Izmir, Menemen, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided